CLINICAL TRIAL: NCT03590418
Title: Intestinal Microbial Diversity of Small Bowel Stoma Effluent and Colonic Feces of Children With Short Bowel Syndrome
Brief Title: Microbial Diversity of Small Bowel Stoma Effluent and Colonic Faeces
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government); National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: ShanghaiXinhua
Record Dates: First submitted 2018-06-15; First posted 2018-07-18 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2017-11

CONDITIONS: Intestinal Failure
Keywords: Intestinal failure; Microbiota
MeSH Terms: conditions — Intestinal Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Intestinal stoma output: No interventions.
- Colonic feaces: No interventions.
- Healthy Control: No interventions.

SUMMARY:
Several studies suggested that dysbacteriosis usually happened in patients with intestinal failure (IF). However, differences of microbiota diversity in small intestine stoma effluents and colonic faeces were rarely studies. Thus this study is aimed to investigate the microbiota compositions and differences of output of small intestine stoma and colon in pediatric IF patients. Fecal samples from IF patients. Each patient received fistula closure in our centre and fecal samples from both small intestinal stoma and colon were collected. Fecal microbial compositions were determined by high-throughput sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intestinal failure. Patients showed good tolerance to parenteral and enteral nutrition administration. Proportion of enteral nutrition is more than 80%.

Stool output maintained at less than 50mL/kg/day. No complications occurred for at least 1 week.

Exclusion Criteria:

* Patients depend mainly on parenteral nutrition. Symptoms like fever, abdominal distention and diarrhea. Complications like parenteral nutrition-associated liver disease, pneumonia and catheter related infection.

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Microbiota diversity and composition clarified by 16s rRNA sequencing | 1)Samples collection: one day before patients are discharged from hospital; 2)DNA extraction: within one week after samples collection; 3)Sequencing and data analyzing: within one month after DNA extract
  DNA of gut microbiota will be extracted. Then purified DNA amplicons are pooled in equimolar and paired-end sequenced (2 × 250) on an Illumina MiSeq platform. Raw Fastq files will be de-multiplexed, quality-filtered using QIIME (version 1.17). Operational taxonomic units (OTUs) will be next clustered with 97% similarity cutoff using UPARSE version 7.1 (http://drive5.com/ uparse/) and chimeric sequences will be identified and removed using UCHIME (http://drive5.com/index.htm). The phylogenetic affiliation of each 16S rRNA gene sequence is analyzed by RDP Classifier (http:// rdp.cme.msu.edu/) against the silva (SSU117/119)16S rRNA. Sobs index and Chao index will be used to evaluate the microbiota diversity. Microbiota composition will be identified on different levels including phylum, family and genus.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xinhua Hospital, affiliated to Shanghai Jiao Tong University, School of Medicine, Shanghai, China

REFERENCES:
- [Background] Arrieta MC, Stiemsma LT, Amenyogbe N, Brown EM, Finlay B. The intestinal microbiome in early life: health and disease. Front Immunol. 2014 Sep 5;5:427. doi: 10.3389/fimmu.2014.00427. eCollection 2014. PMID 25250028
- [Background] Booijink CC, El-Aidy S, Rajilic-Stojanovic M, Heilig HG, Troost FJ, Smidt H, Kleerebezem M, De Vos WM, Zoetendal EG. High temporal and inter-individual variation detected in the human ileal microbiota. Environ Microbiol. 2010 Dec;12(12):3213-27. doi: 10.1111/j.1462-2920.2010.02294.x. PMID 20626454
- [Background] Barrett E, Guinane CM, Ryan CA, Dempsey EM, Murphy BP, O'Toole PW, Fitzgerald GF, Cotter PD, Ross RP, Stanton C. Microbiota diversity and stability of the preterm neonatal ileum and colon of two infants. Microbiologyopen. 2013 Apr;2(2):215-25. doi: 10.1002/mbo3.64. Epub 2013 Jan 24. PMID 23349073
- [Background] Huang Y, Guo F, Li Y, Wang J, Li J. Fecal microbiota signatures of adult patients with different types of short bowel syndrome. J Gastroenterol Hepatol. 2017 Dec;32(12):1949-1957. doi: 10.1111/jgh.13806. PMID 28425133